CLINICAL TRIAL: NCT03366519
Title: Clinical Echography in Emergency Prognostic Evaluation of Pulmonary Embolism: ECU -EP Study.
Acronym: ECU-EP
Status: Withdrawn | Type: Observational
Why Stopped: no open study
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 1608163; 2016-A01721-50 (Other: ANSM)
Record Dates: First submitted 2017-11-21; First posted 2017-12-08 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-03

CONDITIONS: Embolism, Pulmonary
Keywords: Embolism, Pulmonary; echocardiography; emergency; prognosis
MeSH Terms: conditions — Pulmonary Embolism; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with pulmonary embolism: patients with pulmonary embolism confirmed by tomography scan in emergency department
  Interventions: Procedure: clinical echography (CE)

INTERVENTIONS:
Procedure: clinical echography (CE) — clinical echography (CE) is performed in the first 24 hours following the diagnosis of PE, in emergency unit

SUMMARY:
Pulmonary Embolism (PE) is a frequent disease, the third cause of cardiovascular death after stroke and myocardial infarction. According to European guidelines of European Society of Cardiology (ESC) and of European Respiratory Society (ERS), the prognostic stratification of PE severity is mandatory as soon as PE is diagnosed. This stratification includes the hemodynamic status, and specific tools : the assessment of the sPESI score, and the evaluation of PE's impact on right ventricle (RV) : increased biomarkers (troponin, BNP) and right ventricle/left ventricle (RV/LV) ratio.

the RV/LV ration may be evaluated ideally by transthoracic echo (TTE), or by CT scan. Unfortunately, only 10% of patients with PE are evaluated with TTE by a cardiologist in the initial time of PE diagnosis. Hence, the CT scan is the most frequent way to assess RV/LV ratio. However, CT is not possible for all patients (patients with contra-indication) or may have difficulties to provide a clear assessment because of technical issues.

Then, there is a need for morphological evaluation of RV as soon as PE is diagnosed, in every clinical setting. The improvement in technologies allowed the development of clinical echography (CE) in emergency departments.

CE is already available, non-invasive, less expansive, and may be a good way to assess RV/LV ratio in patients with PE diagnosed in emergency departments.

The investigators propose a prospective, multicenter study to assess the sensitivity of CE in patients with PE, compared to CT scan to detect RV/LV ≥0.9.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with pulmonary embolism confirmed
* Simplified Pulmonary Embolism Severity Index (sPESI) ≥ 1

Exclusion Criteria:

* Contra-indication to CT scanner
* Patients with high-risk pulmonary embolism (shock, hypotension)
* Simplified Pulmonary Embolism Severity Index (sPESI) =0

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with a PE confirmed in emergency unit
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-11 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Patients with a measure RV/LV ratio ≥ 0.9 on clinical echography (CE) and CT Scan | day 1
  Sensitivity of clinical echography (CE) to CT Scan to detect an increased RV/LV ratio above 0.9.

SECONDARY OUTCOMES:
Patients with a measure RV/LV ratio < 0.9 on clinical echography (CE) and CT Scan | day 1
  Specificity of clinical echography (CE) to CT Scan to detect an increased RV/LV ratio below 0.9
Patients with abnormal inferior vena cava. | day 30
death | day 30

CONTACTS AND LOCATIONS:
Overall Officials: Alain Viallon, MD PhD, Principal Investigator — Centre Hospitalier Universitaire de Saint Etienne

IPD SHARING:
Plan to Share IPD: No